CLINICAL TRIAL: NCT04583657
Title: To Evaluate the Intestinal Tolerance and Health Effects of Daily Consumption of Two Eggs With a Particular Fatty Acid Profile on a Set of Parameters Related to Metabolic Disorders
Brief Title: Intestinal Tolerance & Health Effects of Daily Consumption of Two Eggs With Fatty Acid Profile Related to Metabolic Disorders
Acronym: Oil4Egg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Oil4Egg
Record Dates: First submitted 2020-09-03; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Healthy; Abdominal Obesity; Sedentary Behavior
MeSH Terms: conditions — Obesity, Abdominal; Sedentary Behavior | interventions — Eggs

STUDY DESIGN:
Intervention Model Description: This monocentric study is an interventional, randomized, double-blind, controlled study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Consumption of two "classical eggs" per day during three months. The fatty acid pattern of those eggs is characterized by: total saturated fatty acid 34.25%, total monounsaturated fatty acid 47.68%, total n-6 polyunsaturated fatty acid 16.97%, total n-3 polyunsaturated fatty acid 1.10%.
  Interventions: Other: Eggs
- Test (Experimental): Consumption of two test eggs per day during three months. These eggs are naturally enriched in n-3 polyunsaturated fatty acids, conjugated-linoleic acids and conjugated-linolenic acids (total saturated fatty acid 31.74%, total monounsaturated fatty acid 28.09%, total n-6 polyunsaturated fatty acid 16.07%, total n-3 polyunsaturated fatty acid 6.51%)
  Interventions: Other: Eggs

INTERVENTIONS:
Other: Eggs — Consumption of two eggs (control or test) per day during three months

SUMMARY:
This study has two objectives: 1) to check that the daily consumption of two eggs with a particular fatty acid pattern rich in n-3 polyunsaturated fatty acids (α-linolenic acid, docosahexaenoic acid), conjugated-linoleic acid and conjugated-linolenic acid is well tolerated by the consumer ; 2) to evaluate the effects of the consumption of these eggs on health parameters in subjects presenting a risk of developing a metabolic disorder.

This monocentric study is an interventional, randomized, double-blind, control study.

DETAILED DESCRIPTION:
n-3 polyunsaturated fatty acids, conjugated-linoleic acids and conjugated-linolenic acids show interesting effects in the context of health. Indeed, some studies suggest positive effects on circulating lipids or inflammation associated with certain disorders such as diabetes, following the consumption of these fatty acids.

However, these fatty acids are not very present in the classic diet. Therefore, we have developped hens eggs naturally enriched in n-3 polyunsaturated fatty acids, conjugated-linoleic acids and conjugated-linolenic acids by changing the hens feed.

This study has two objectives: 1) to check that the daily consumption of two eggs with a particular fatty acid pattern rich in n-3 polyunsaturated fatty acids (α-linolenic acid, docosahexaenoic acid), conjugated-linoleic acid and conjugated-linolenic acid is well tolerated by the consumer ; 2) to evaluate the effects of the consumption of these eggs on health parameters in subjects presenting a risk of developing a metabolic disorder.

To do this, 80 subjects aged 35 to 75, sedentary (<2 hours of physical activity per week) and with abdominal obesity (> 94cm for men and> 80cm for women) were recruited and were divided into two groups: the control group (12 subjects consuming 2 classic eggs for 3 months per day) or the test group (12 subjects consuming 2 eggs enriched in omega per day for 3 months).

A medical examination with blood sampling was scheduled every month at baseline (Day 0), after one month (Day 30), after two months (Day 60) and at the end of the 3 months of intervention (Day90). During those visits, the following were monitored: glucose parameters, lipids parameters, fatty acid profile of red blood cells and plasma and safety parameters related to haematology, kidney and liver functions .

During these monthly medical visits patients also completed the questionnaires assessing intestinal tolerance (visual analogue scale showing 10 gastrointestinal symptoms), satiety (visual analog scale questionnaire) and well-being (36 items short form survey). Eating habits were monitored using a food diary. Additional parameters were measured only during the first and the last visit: coagulation, nutritional status, endothelial function and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Woman or man, aged of 35 to 75 years
* Abdominal obesity : waist circumference for men > 94cm and > 80cm for women
* Practicing < 2h of physical activity per week

Exclusion Criteria:

* Uncontrolled systolic blood pressure > 160/100mmHg
* For premenopausal women: pregnant or lactating women
* For menopausal women: less than 6 months of menopause
* Perimenopausal women with symptoms
* Type II diabetes (fasted glycaemia ≥ 126mg/dl or HbA1c ≥ 6.5%), Type I diabetes
* Medical history or actual cardiovascular disease (myocardial infarction, angina, transient ischemic attack, lower limb arteriopathy)
* Familial history of premature cardiovascular incident (in male first degree relative < 55 years and in female first degree relative < 65 years; myocardial infarction, angina, transient ischemic attack, lower limb arteriopathy)
* Medical history or actual liver, pancreas, kidney, pulmonary or gastrointestinal problem
* Thyroid disorder
* Cancer < 5 years before the screening visit
* Smokers or who have stopped smoking within 6 months before the screening visit
* Subject presenting allergy or food intolerance to eggs
* Subjects with psychiatric problems and/or using antipsychotics
* Drug addiction problem
* Recent change of body weight > 5kg (< 3 months before the screening visit)
* Within 3 months before the screening visit, change in the chronic (> 7 days in a row) intake or dosage of drug(s) or product(s) modifying

  * The glucose or lipid metabolism
  * The blood pressure and heart rate
  * Intestinal tolerance
  * Hepatic, pancreas or kidney functions
  * Satiety
  * The inflammatory status
* Current or recent (< 3 months before the screening visit) intake of dietary supplements rich in n-3 polyunsaturated fatty acid
* Vegan diet
* Consumption of fish > 3 times per week
* Subjects who drink more than 3 glasses of alcohol per day (> 30 g of alcohol per day)
* LDL > 159 mg/dl or total cholesterol > 239 mg/dl or triglyceride > 200 mg/dl or HDL < 40 mg/dl
* Docosahexaenoic acid in red blood cell phospholipids > 8 %
* Subjects having participated to another clinical trial < 1 month before the screening test visit

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Glycated haemoglobin (HbA1c) | Change from baseline (visit 1) glycated haemoglobin at 3 months (Day 90, visit 4)
  Glycated haemoglobin (HbA1c) in blood samples

SECONDARY OUTCOMES:
Glucose | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Insulin | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Homeostatic model assessment (HOMA) | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Quantitative insulin sensitivity check index (QUICKI) | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Triglycerides | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Total cholesterol | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
low-density lipoprotein (LDL) cholesterol | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
high-density lipoprotein (HDL) cholesterol | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
non-high-density lipoprotein cholesterol (non-HDL) | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Fatty acid pattern in red blood cells | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Fatty acid pattern plasma | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Urea | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Uric acid | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Creatinine | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Glomerular filtration rate (GFR) | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Sodium (Na) | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Potassium (K) | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Chlore (Cl) | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Phosphate (P) | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Alanine transaminase (ALAT) | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Aspartate aminotransferase (ASAT) | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Gamma-glutamyl transferase (GGT) | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Alkaline phosphatase (ALP) | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Lipase | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Haemoglobin | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Mean corpuscular volume (MCV) | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Mean corpuscular hemoglobin concentration (MCHC) | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Red blood cells | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
White blood cells | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Blood cell count | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Reticulocytes | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Haematocrit | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  blood samples
Body weight | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  Impedancemeter
Waist circumference | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  Measuring tape
Hip circumference | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  Measuring tape
Fat mass | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  Impedancemeter
Lean mass | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  Impedancemeter
Visceral fat mass | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  Impedancemeter
International normalized ratio (INR) | baseline (visit 1) and Day 90 (last visit 4)
  blood samples
Activated clotting time (ACT) | baseline (visit 1) and Day 90 (last visit 4)
  blood samples
Iron | baseline (visit 1) and Day 90 (last visit 4)
  blood samples
Transferrin | baseline (visit 1) and Day 90 (last visit 4)
  blood samples
Ferritin | baseline (visit 1) and Day 90 (last visit 4)
  blood samples
% transferrin saturation | baseline (visit 1) and Day 90 (last visit 4)
  blood samples
Vitamin B12 | baseline (visit 1) and Day 90 (last visit 4)
  blood samples
25-hydroxy-vitamin D | baseline (visit 1) and Day 90 (last visit 4)
  blood samples
Protein | baseline (visit 1) and Day 90 (last visit 4)
  blood samples
Albumin | baseline (visit 1) and Day 90 (last visit 4)
  blood samples
C-reactive protein (CRP) | baseline (visit 1) and Day 90 (last visit 4)
  blood samples
Interleukin-6 | baseline (visit 1) and Day 90 (last visit 4)
  blood samples
Interleukin-1b | baseline (visit 1) and Day 90 (last visit 4)
  blood samples
Tumor necrosis factor alpha (TNFa) | baseline (visit 1) and Day 90 (last visit 4)
  blood samples
Oxidized low-density lipoprotein (LDLox) | baseline (visit 1) and Day 90 (last visit 4)
  blood samples
Nitrosylated hemoglobin (HbNO) | baseline (visit 1) and Day 90 (last visit 4)
  blood samples
Satiety | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  visual analog scale questionnaire
Intestinal tolerance | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  visual analog scale questionnaire
Quality of life 36-item short-form survey (SF36) | baseline (visit 1), Day 30 (visit 2), Day 60 (visit 3) and Day 90 (last visit 4)
  SF36 questionnaire
Reactive hyperemia index (LnRHI) | baseline (visit 1) and Day 90 (last visit 4)
  Tonometry
Augmentation index normalized for heart rate (AI@75bpm) | baseline (visit 1) and Day 90 (last visit 4)
  Tonometry
Systolic blood pressure | baseline (visit 1) and Day 90 (last visit 4)
  Tensiometer
Diastolic blood pressure | baseline (visit 1) and Day 90 (last visit 4)
  Tensiometer
Glycated haemoglobin (HbA1c) | Day 30 (visit 2) and Day 60 (visit 3)
  Glycated haemoglobin in blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Yvan Larondelle, Prof, Study Director — Université Catholique de Louvain
Locations (1):
- Center of Investigation in Clinical Nutrition, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No